CLINICAL TRIAL: NCT03651076
Title: Randomized Controlled Trial of Panniculus Retraction Methods for Cesarean Delivery
Brief Title: Traxi Panniculus Retractor for Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual due to provider preference
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Clinical Innovations, LLC (Industry); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ai-ris Collier, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P000369
Record Dates: First submitted 2018-07-18; First posted 2018-08-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Morbid; Cesarean Section Complications
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Traxi panniculus retraction group (Experimental): The method of panniculus retraction will be the Traxi panniculus retraction (Clinical Innovations, LLC) by the provider.
  Interventions: Device: Traxi panniculus retraction (Clinical Innovations, LLC)
- Standard of care (No Intervention): Standard methods of panniculus retraction as determined by individual provider (including medical taping, extra personnel for retraction)

INTERVENTIONS:
Device: Traxi panniculus retraction (Clinical Innovations, LLC) — class I, FDA-exempt, commercially available for use in panniculus retraction during cesarean delivery or other laparotomy
  Arms: Traxi panniculus retraction group

SUMMARY:
This prospective, open-label, randomized-controlled trial is designed to evaluate the use of the Traxi panniculus retractor-- a commercially available Class I FDA-exempt device will improve surgical outcomes, cardiopulmonary function, and provider/patient satisfaction in morbidly obese women undergoing cesarean delivery.

DETAILED DESCRIPTION:
Morbidly obese women (BMI >/= 40) undergoing non-emergent cesarean delivery will be recruited and randomized to Traxi panniculus retraction or standard of care for panniculus retraction.

The primary outcome evaluated will be operating time (incision to closure). Other secondary outcomes related to surgery including estimated blood loss, surgical site infection, and number of scrubbed personnel.

A secondary aim of the study is to evaluate the hypothesis that the Traxi retraction device reduces chestwall compression panniculus retraction and will improve intraoperative pulmonary function. To do this, the investigators will measure the difference in individual participant pulmonary function tests (forced vital capacity, forced expiratory volume) before and after panniculus retraction using a bedside spirometer.

A tertiary aim of the study is to evaluate the hypothesis that the Traxi retraction device will improve patient and provider satisfaction due to improved delivery experience and maintaining patient dignity. Patient and provider-reported outcomes will be evaluated using surveys.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* BMI greater than or equal to 40 kg/m^2
* Undergoing non-emergent cesarean delivery
* Able and willing to provide written, informed consent
* Singleton gestation

Exclusion Criteria:

* Fetal demise
* Disruption of abdominal skin (infection, rash, abrasion, laceration)
* Known adhesive allergy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Cesarean delivery operative time | through study completion, approximately 6 to 8 weeks
  time from skin incision to closure during cesarean delivery

SECONDARY OUTCOMES:
Change in pulmonary function (forced vital capacity) | through study completion, approximately 6 to 8 weeks
  measure difference in pulmonary function tests (FVC=forced vital capacity) before and after application of panniculus retraction method
Change in pulmonary function (forced expiratory volume) | through study completion, approximately 6 to 8 weeks
  measure difference in pulmonary function tests (FEV1=forced expiratory volume in 1 minute) before and after application of panniculus retraction method
Patient satisfaction assessed by a questionnaire | through study completion, approximately 6 to 8 weeks
  patient-reported outcomes regarding surgery and delivery will be obtained using a survey made by the research team with a four level likert scale
Provider satisfaction with a survey | through study completion, approximately 6 to 8 weeks
  provider-reported outcomes regarding surgery will be obtained using survey with an eleven level likert scale

OTHER OUTCOMES:
Estimated blood loss | through study completion, approximately 6 to 8 weeks
  estimated blood loss reported on operative report
Wound complication | through study completion, approximately 6 to 8 weeks
  review of medical records for 6 weeks postpartum to evaluate for wound opening or infection rates
Number of personnel involved in cesarean | through study completion, approximately 6 to 8 weeks
  recorded number of scrubbed personnel needed to assist with surgery
Hospital length of stay | through study completion, approximately 6 to 8 weeks
  inpatient length of stay post-delivery
Composite neonatal outcome | through study completion, approximately 6 to 8 weeks
  composite rate of neonatal intensive care unit (NICU) admission, 5-minute Apgar score <7)

CONTACTS AND LOCATIONS:
Overall Officials: Ai-ris Collier, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT03651076/Prot_SAP_ICF_000.pdf